CLINICAL TRIAL: NCT00038532
Title: An Open Label, Phase II Study of Amprenavir/Ritonavir, Saquinavir/Ritonavir or Efavirenz in HIV-Infected Subjects Following Failure With Kaletra (ABT-378/Ritonavir) as Their First Protease Inhibitor Based HAART
Brief Title: Amprenavir/Ritonavir, Saquinavir/Ritonavir or Efavirenz in HIV-Infected Subjects Following Failure With Kaletra (ABT-378/Ritonavir) as Their First Protease Inhibitor Based HAART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M01-287; NCT00021619 (obsolete NCT alias)
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: treatment experienced; HIV
MeSH Terms: conditions — HIV Infections | interventions — amprenavir; Ritonavir; Saquinavir; efavirenz

INTERVENTIONS:
Drug: Amprenavir/ritonavir
Drug: Saquinavir/ritonavir
Drug: Efavirenz

SUMMARY:
The purpose of this study is to study amprenavir/ritonavir, saquinavir/ritonavir or efavirenz in HIV-infected patients following failure with Kaletra (ABT-378/ritonavir) as their first protease inhibitor based HAART.

ELIGIBILITY:
Inclusion:

* Remain on present anti-HIV drugs during screening until a new regimen is started.
* Have a viral load of at least 1,000 copies/ml on the 2 most recent tests after at least 24 weeks of lopinavir/ritonavir and while still on it.
* Have an HIV which shows reduced susceptibility to lopinavir.
* Are at least 18 years old.
* Are not presently ill.
* Have not been treated for an opportunistic infection within 30 days of screening.
* Agree not to take certain drugs and agree to inform and get permission from the doctor before taking any medicines, over the counter medicines, herbal medicines, alcohol or recreational drugs.
* Agree to use an accepted barrier method of birth control.

Exclusion:

* Female subject is pregnant or lactating.
* Have taken any protease inhibitor other than lopinavir/ritonavir for more that two weeks.
* Are taking chemotherapy.
* Have a medical problem with their pancreas.
* Have been screened for this study within the past 12 weeks.
* Appear to be unsuitable in the opinion of the doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2001-04

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV RNA levels below the limit of quantification (400 copies/mL) at week 24 and the time until loss of virologic response through week 48

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sun, M.D., Study Chair — Divisional Vice President, Infectious Diseases and Virology Development
Locations (54):
- United States (26):
  - Phoenix Body Positive, Inc., Phoenix, Arizona
  - Paul J. Cimoch, M.D., Fountain Valley, California
  - AIDS Health Care Foundation - Research Center, Los Angeles, California
  - Tower Infectious Diseases Medical Associates, Los Angeles, California
  - 20th Avenue Medical Center Kaiser Permanente, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - IDC Research Initiative, Altamonte Springs, Florida
  - Gary J. Richmond, M.D., Fort Lauderdale, Florida
  - Associates in Research, Fort Myers, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Infectious Disease Research Institute, Inc., Tampa, Florida
  - AIDS Research Consortium of Atlanta, Inc., Atlanta, Georgia
  - CORE Center, Chicago, Illinois
  - Donna E. Sweet, M.D., Wichita, Kansas
  - David Parks, M.D., St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - Howard A. Grossman, M.D., New York, New York
  - John B. Montana, M.D., New York, New York
  - State University of New York at Stony Brook, Stony Brook, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Research & Education Group, Portland, Oregon
  - Bornemann Internal Medicine, Reading, Pennsylvania
  - David Wright, M.D., Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Diversified Medical Practices, P.A., Houston, Texas
  - Hampton Roads Medical Specialists, Hampton, Virginia
- Argentina (2):
  - Hospital Muniz - FUNDAI, Buenos Aires
  - Fundacion Huesped, Buenos Aires
- Hospital Heliopolis, São Paulo, Brazil
- Canada (3):
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Toronto General Hospital Division of The University Health Network, Toronto, Ontario
  - Montreal Chest Institute/Royal Victoria Hospital, Montreal, Quebec
- France (6):
  - Hopital Michalon - C.H.U. de Grenoble, Grenoble
  - Groupe Hospitalier Cochin -Saint-Vincent-de-Paul La Roche-Guyon, Paris
  - Hopital Tenon, Paris
  - Hospital Yves Le Foll, Saint-Brieuc
  - La Seyne sur Mer, Hopital Chalucet, Toulon
  - C.H.U. Brabois - Tour Drouet, Rue du Morvan, Vandœuvre-lès-Nancy
- Germany (5):
  - CORE Center, Berlin
  - Universitatsklinikum, Düsseldorf
  - Klinikum J.W. Goethe Universitat, Frankfurt
  - Institut fur Immunologie Pathologie und Molekularbiologie, Hamburg
  - Albrecht Ulmer, M.D., Stuttgart
- S. Raffaele Hospital, Milan, Italy
- Wojewodzki Szpital Zakazny, Warsaw, Poland
- Puerto Rico (2):
  - Centro Familiar, Inc, Ponce
  - New Puerto Rico CONCRA, Rio Piedras
- Spain (6):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital De La Sta Creu I San Pau, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Carlos III, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Vergen del Rocio, Seville
- Royal Free Hospital, London, United Kingdom